CLINICAL TRIAL: NCT05757986
Title: Dynamic Predictive Model for Postoperative Nausea and Vomiting for Patient Received Gynecological Laparoscopic Surgery
Brief Title: Predictive Model for PONV for Patient Received Gynecological Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiang Liu (Other)
Responsible Party: Sponsor-Investigator, Jiang Liu, Principal Investigator, Weifang Medical University
Organization: Weifang Medical University (Other)
Other Study IDs: 2023YX030
Record Dates: First submitted 2023-02-22; First posted 2023-03-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group
  Interventions: Other: The presence of nausea and vomiting within 24 hours after surgery
- Control group
  Interventions: Other: The presence of nausea and vomiting within 24 hours after surgery

INTERVENTIONS:
Other: The presence of nausea and vomiting within 24 hours after surgery — This is a prospective risk prediction model building, thus there is no traditional definition of intervention.

SUMMARY:
This is a prospective study to dynamically predict the risk of PONV in patients undergoing gynecologic laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

-All female patients receiving gynecological laparoscopic surgery.

Exclusion Criteria:

-Patients requiring intraoperative open-surgery, requiring other procedures in addition to gynecological laparoscopy, with severe organ dysfunction, unstable postoperative vital signs or requiring transfer to ICU.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The objective of this study was to develop a risk prediction model for postoperative nausea and vomiting in patients undergoing gynecologic laparoscopic surgery. Therefore, the target population of this study was limited to female patients with gynecologic diseases and requiring gynecologic laparoscopic surgery.
Study Population: The female patients with gynecological diseases and requiring gynecological laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
PONV | Within 24 hours after surgery
  The occurrence and severity of PONV is evaluated by Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Weifang Medical University, Weifang, Shangdong, China